CLINICAL TRIAL: NCT05001776
Title: Choice of the Optimal Method for Treatment of Acute Thrombophlebitis of the Varicose Great Saphenous Vein: Comparison of Endovenous Laser Ablation and Conservative Approach
Brief Title: Endovenous Laser Ablation in Acute Thrombophlebitis of the Varicose Great Saphenous Vein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-06/21
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Superficial Vein Thrombosis; Endovenous Laser Ablation
Keywords: acute thrombophlebitis; acute thrombosis; superficial vein of leg; great saphenous vein; various vein; endovenous laser ablation; fondaparinux
MeSH Terms: interventions — Fondaparinux

STUDY DESIGN:
Intervention Model Description: Prospective single-centre open-label randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endovenous laser ablation without anticoagulants (Active Comparator): Endovenous laser ablation without using of any anticoagulant
  Interventions: Procedure: Endovenous laser ablation
- Endovenous laser ablation with short-term anticoagulant (Active Comparator): Endovenous laser ablation and subsequent 7 days of subcutaneous fondaparinux sodium
  Interventions: Procedure: Endovenous laser ablation; Drug: Fondaparinux Sodium
- Medical treatment (Active Comparator): 45 days of subcutaneous fondaparinux sodium
  Interventions: Drug: Fondaparinux Sodium

INTERVENTIONS:
Procedure: Endovenous laser ablation — Laser ablation of the great saphenous vein close to sapheno-femoral junction
  Other Names: Ablation of varicose vein
  Arms: Endovenous laser ablation with short-term anticoagulant; Endovenous laser ablation without anticoagulants
Drug: Fondaparinux Sodium — Fondaparinux sodium for 7 days or 45 days
  Other Names: Anticoagulation
  Arms: Endovenous laser ablation with short-term anticoagulant; Medical treatment

SUMMARY:
Рrospective single-centre randomized open-label study for comparison three modes of treatment for thrombosis of varicose great saphena vein - standard medical with fondaparinux sodium for 45 days, endovenous laser ablation close to the saphenofemoral junction with a 7-day course of anticoagulation and endovenous laser ablation close to the saphenofemoral junction without the use of anticoagulants.

DETAILED DESCRIPTION:
Superficial venous thrombosis is a common complication in patients with varicose veins of low extremities. The most dangerous consequence of such thrombosis is its propagation to deep veins and subsequent pulmonary embolism. Recommended mode of treatment for superficial vein thrombosis is a prolonged usage of anticoagulants (preferably fondaparinux sodium for least 45 days as the best-studied approach). However, it may be not suitable for some patients, for example with a high risk of bleeding. Another possible mode of treatment is endovenous laser ablation of the saphenous vein very close to the saphenofemoral junction. This a minimally invasive procedure that may be performed ambulatory is able to decrease the risk of deep veins thrombosis and possibly allow to shorten or even eliminate the necessity of anticoagulant use. Such a suggestion was not appropriately studied in randomized clinical trials.

The aim of this prospective single-centre randomized open-label study is to compare three modes of treatment for thrombosis of varicose great saphena vein - standard medical with fondaparinux sodium, endovenous laser ablation close to the saphenofemoral junction with shortening the course of anticoagulation and endovenous laser ablation close to the saphenofemoral junction without the use of anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Acute thrombosis of varicose great saphenous vein and/or its major branches more than 5 cm from the saphenofemoral junction
* Signed informed consent

Exclusion Criteria:

* More than 3 weeks after symptom onset
* Ultrasound signs of deep vein thrombosis
* Suspected pulmonary embolism
* Superficial vein thrombosis within 5 cm from the saphenofemoral junction
* Bilateral superficial vein thrombosis
* Thrombosis of subfascial part of perforating veins to the level of fascia
* Thrombosis of small saphenous vein
* Superficial vein thrombosis associated with sclerotherapy
* History of deep vein thrombosis and/or pulmonary embolism
* Superficial vein thrombosis within 3 months before inclusion
* Anemia (haemoglobin less than 90 g/l)
* Low platelet count (less than 100 X 109/l)
* Severe renal impairment (calculated GFR less than 20 ml/min/1,73 m2)
* Body mass less than 50 kg
* Morbid obesity (BMI higher than 40 kg/m2)
* Allergy to fondaparinux sodium and local anaesthetics
* Using anticoagulants for treating the current episode of venous thrombosis
* Using anticoagulants for other medical conditions (e.g. atrial fibrillation)
* Double antiplatelet therapy
* Regular use of NSAIDs (except aspirin less than 325 mg daily)
* High risk of bleeding according to an investigator
* Active clinically relevant bleeding
* Clinically relevant bleeding within last 30 days before inclusion
* Major surgery of severe head trauma within last 30 days before inclusion
* Ophthalmic, spinal or cerebral surgery within last 12 months
* Active gastric or duodenum ulcer, erosive and ulcerative gastrointestinal disorder
* Documented haemorrhagic diathesis
* Uncontrolled arterial hypertension (systolic[180 mm Hg, diastolic[110 mm Hg)
* Active cancer, history of cancer
* Acute illness, decompensation of chronic illness
* Autoimmune disease, treatment of autoimmune disease
* Severe chronic heart failure and/or marked oedema due to heart failure
* Severe pulmonary insufficiency
* Bacterial endocarditis
* Severe renal failure
* Known severe thrombophilia (antiphospholipid syndrome, a deficit of antithrombin, a deficit of protein C, S, factor V Leiden, prothrombin G20210A)
* Immobility, unable to increase mobility
* Pregnant or breastfeeding women
* Alcohol abuse, drugs abuse or other circumstances indication low compliance
* Unwilling of unable to follow requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Composite of deep vein thrombosis, symptomatic pulmonary embolism, superficial vein thrombosis extension, superficial vein thrombosis recurrence or thrombosis of subfascial part of perforating veins to the level of fascia | 45 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Major bleedings | 45 days
  Major bleedings according to ISTH definition

SECONDARY OUTCOMES:
Composite of deep vein thrombosis, symptomatic pulmonary embolism, superficial vein thrombosis extension, superficial vein thrombosis recurrence or thrombosis of subfascial part of perforating veins to the level of fascia | 7 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Composite of deep vein thrombosis, symptomatic pulmonary embolism, superficial vein thrombosis extension, superficial vein thrombosis recurrence or thrombosis of subfascial part of perforating veins to the level of fascia | 90 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Composite of death, symptomatic deep vein thrombosis, symptomatic pulmonary embolism, symptomatic superficial vein thrombosis extension or symptomatic superficial vein thrombosis recurrence | 7 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Composite of death, symptomatic deep vein thrombosis, symptomatic pulmonary embolism, symptomatic superficial vein thrombosis extension or symptomatic superficial vein thrombosis recurrence | 45 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Composite of death, symptomatic deep vein thrombosis, symptomatic pulmonary embolism, symptomatic superficial vein thrombosis extension or symptomatic superficial vein thrombosis recurrence | 90 days
  All vein thrombosis should be confirmed by ultrasonography, pulmonary embolism - by computed tomography. Supreficial vein thrombosis extension - increasing size of existing thrombosis at least 2 cm. Superficial vein thrombosis recurrence - thrombosis of new superficial vein not related to index thrombosis or new thrombosis in the same superficial vein clearly separated from index thrombosis by segment on vein without signs of thrombosis at least 10 cm in length
Major bleedings | 7 days
  Major bleedings according to ISTH definition
Major bleedings | 90 days
  Major bleedings according to ISTH definition
All bleedings | 7 days
  All overt bleedings classified as major, clinically relevant non-major and minor according to ISTH criteria
All bleedings | 45 days
  All overt bleedings classified as major, clinically relevant non-major and minor according to ISTH criteria
All bleedings | 90 days
  All overt bleedings classified as major, clinically relevant non-major and minor
Bleedings according to BARC criteria | 7 days
  Overt bleedings classified with BARC criteria
Bleedings according to BARC criteria | Overt bleedings classified with BARC criteria
  Overt bleedings classified with BARC criteria
Bleedings according to BARC criteria | 90 days
  Overt bleedings classified with BARC criteria

OTHER OUTCOMES:
Surgical intervention for superficial vein thrombosis | 45 days
  Requirement of unplanned surgical intervention for treatment of superficial vein thrombosis
Surgical intervention for superficial vein thrombosis | 90 days
  Requirement of unplanned surgical intervention for treatment of superficial vein thrombosis
Severity of pain | 7 days
  10 cm visual analog scale of pain and 0-10 numeric pain rating score (0 - no pain, 10 - worst imaginable pain)
Severity of pain | 45 days
  10 cm visual analog scale of pain and 0-10 numeric pain rating score (0 - no pain, 10 - worst imaginable pain)
Severity of pain | 90 days
  10 cm visual analog scale of pain and 0-10 numeric pain rating score (0 - no pain, 10 - worst imaginable pain)
Quality of life according to 36-Item Short Form Health Status Survey | 7 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability
Quality of life according to 36-Item Short Form Health Status Survey | 45 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability
Quality of life according to 36-Item Short Form Health Status Survey | 90 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability
Quality of life according to European Quality of Life Questionnaire EQ-5D-3L | 7 days
  Zero score is equivalent to no disability and a score of 10 is equivalent to maximal disability
Quality of life according to European Quality of Life Questionnaire EQ-5D-3L | 45 days
  Zero score is equivalent to no disability and a score of 10 is equivalent to maximal disability
Quality of life according to European Quality of Life Questionnaire EQ-5D-3L | 90 days
  Zero score is equivalent to no disability and a score of 10 is equivalent to maximal disability
Quality of life according to Chronic Venous Disease quality of life Questionnaire (CIVIQ-20) | 7 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability
Quality of life according to Chronic Venous Disease quality of life Questionnaire (CIVIQ-20) | 45 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability
Quality of life according to Chronic Venous Disease quality of life Questionnaire (CIVIQ-20) | 90 days
  Zero score is equivalent to maximum disability and a score of 100 is equivalent to no disability

CONTACTS AND LOCATIONS:
Overall Officials: Igor S Yavelov, MD, Principal Investigator — National Medical Research Center for Therapy and Preventive Medicine
Locations (1):
- National Medical Research Center for Therapy and Preventive Medicinel, Moscow, Russia